CLINICAL TRIAL: NCT07200479
Title: A Clinical Study to Explore the Safety, Efficacy and Cellular Metabolic Kinetics of CT1194D CAR-T Cells Injection in Patients With Relapsed/Refractory B-Cell Neoplasms
Brief Title: A Clinical Study to Explore CT1194D in Patients With Relapsed/Refractory B-Cell Neoplasms
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025099
Record Dates: First submitted 2025-09-19; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory B-Cell Neoplasms
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells chimeric antigen receptor T cells (Experimental)
  Interventions: Drug: CAR T cells chimeric antigen receptor cells

INTERVENTIONS:
Drug: CAR T cells chimeric antigen receptor cells — CT1194D cells infusion

SUMMARY:
A Clinical Study to Explore the Safety, Efficacy and Cellular Metabolic Kinetics of CT1194D CAR-T Cells Injection in Patients with Relapsed/Refractory B-Cell Neoplasms

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose exploratory clinical study to evaluate the safety, efficacy, cellular Metabolic Kinetics of CT1194D CAR-T Cells in patients with relapsed/refractory B-cell Non-Hodgkin's Lymphoma (R/R B-NHL) and relapsed/refractory B-cell acute lymphoblastic leukemia (R/R B-ALL). It is planned to enroll around 20-30 participants.

ELIGIBILITY:
Inclusion Criteria:

* R/R B-NHL Inclusion Criteria：

  1. Voluntary participation in the clinical study; I fully understand and are informed of this study and sign the informed consent form; Willing to follow and able to complete all study procedures; 2. Age 18-75 years (inclusive) 3. Histologically or cytologically confirmed diagnosis of R/R B-NHL according to the WHO classification of lymphoid hyperplasia and neoplasms, 5th Edition 2022, including:

  1) Cohort A1: large B-cell lymphoma, including diffuse large B-cell lymphoma unspecified (DLBCL, NOS), primary mediastinal large B-cell lymphoma (PMBCL), high-grade B-cell lymphoma, large B-cell lymphoma transformed from follicular lymphoma (FLBL)/Grade 3b FL; 2) Cohort A2: Mantle cell lymphoma (MCL); 3) Cohort B: follicular lymphoma grade 1-3a; 4. Prior Therapy Requirements:
  1. Cohort A1: Patients who have previously received standard systemic therapy, including regimens containing anti-CD20 drugs (except CD20 negative) and anthracyclines;
  2. Cohort A2: Prior standard systemic therapy, including an anti-CD20 agent (except CD20 negative), an anthracycline-containing regimen, or a BTK inhibitor;
  3. Cohort B: previously received standard systemic therapy, including regimens containing anti-CD20 drugs (except CD20 negative) and anthracyclines; 5. Intolerance during the last treatment, or the need for new treatment after the last adequate treatment (at least 2 cycles) or as assessed by the investigator; 6. At least one of the following:

  1) As measured by CT: Nodal lesions > 1.5 cm in long diameter or extranodal lesions > 1.0 cm in long diameter and measurable in short axis; 2) As measured by PET: FDG uptake fraction of 4 or 5; 8. Eastern Cooperative Oncology Group (ECOG) score 0-1; 9. Participants should meet the following test results (there should be no ongoing supportive care):
  1. Hematology: ① Platelet (PLT) ≥ 75 × 109/L (study participants with bone marrow or peripheral blood involvement: PLT ≥ 50 × 109/L), ② Hemoglobin (Hb) ≥ 80 g/L (study participants with bone marrow or peripheral blood involvement: Hb ≥ 60 g/L);
  2. Endogenous creatinine clearance ≥ 50 mL/min, or creatinine ≤ 1.5 × ULN (using Cockcroft-Gault formula);
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN, total bilirubin ≤ 1.5 × ULN; If lymphoma invades the liver: AST and ALT ≤ 5 × ULN, total bilirubin ≤ 3.0 × ULN;
  4. International normalized ratio (INR) and activated partial thromboplastin time (APTT) were required to be ≤ 1.5 × ULN.
  5. Oxygen saturation ≥ 92% in non-oxygen inhalation state;
  6. Left ventricular ejection fraction (LVEF) ≥ 50% (LVEF value near the cut-off value can be enrolled after adequate risk assessment by the investigator); 10. Female participants of child-bearing potential must have a negative pregnancy test at the time of screening and before receiving lymphodepletion therapy, be willing to use a highly effective and reliable method of contraception within 1 year after receiving study treatment, and absolutely prohibit egg donation within 1 year after receiving study treatment infusion during the study; A male participant, if sexually active with a female of childbearing potential, is willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment. All male participants absolutely refrain from donating sperm for 1 year after receiving study treatment infusion during the study.
* R/R B-ALL Inclusion Criteria：

  1. Voluntary participation in the clinical study; I fully understand and are informed of this study and sign the informed consent form; Willing to follow and able to complete all study procedures;
  2. Age 18-75 years (inclusive);
  3. Morphologically, immunologically, or molecularly confirmed diagnosis of R/R B-ALL (Cohort C) and 1 of the following criteria is met:

  <!-- -->

  1. Patients who did not achieve complete remission after standard induction regimen chemotherapy or had early relapse after complete remission (< 12 months) or late relapse after complete remission (≥ 12 months) and did not achieve complete remission after standard one course of induction regimen chemotherapy and relapsed after 2 or more CR or CRi;
  2. For Ph + ALL patients who have not achieved complete remission after receiving at least one TKI treatment in addition to standard induction chemotherapy, or relapsed after complete remission (those who cannot tolerate TKI treatment or have contraindications for TKI treatment, or have T315I mutation are not required to receive TKI treatment); 4. Leukemia cells with positive expression of CD19 and/or CD20 in bone marrow or peripheral blood; 5. Bone marrow cell morphology or peripheral blood indicates blast ratio ≥ 5%; 6. Estimated survival > 12 weeks; 7. Eastern Cooperative Oncology Group (ECOG) score 0-2; 8. Participants should meet the following test results (there should be no ongoing supportive care):

  <!-- -->

  1. Endogenous creatinine clearance ≥ 50 mL/min, or creatinine ≤ 1.5 × ULN (using the Cockcroft-Gault formula);
  2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN, total bilirubin ≤ 1.5 × ULN; If hepatobiliary involvement: AST and ALT ≤ 5 × ULN, total bilirubin ≤ 3.0 × ULN;
  3. International normalized ratio (INR) and activated partial thromboplastin time (APTT) must be ≤ 1.5 × ULN;
  4. Oxygen saturation ≥ 92% in non-oxygen inhalation state;
  5. Left ventricular ejection fraction (LVEF) ≥ 50% (LVEF values near the cut-off value may be enrolled after adequate risk assessment by the investigator).

  9. Female participants of child-bearing potential must have a negative pregnancy test at the time of screening and before receiving lymphodepletion therapy, be willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment, and absolutely refrain from egg donation for 1 year after receiving study treatment infusion during the study; A male participant, if sexually active with a female of childbearing potential, is willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment. All male participants absolutely refrain from donating sperm for 1 year after receiving study treatment infusion during the study.

Exclusion Criteria:

* R/R B-NHL Exclusion Criteria：

  1. Pregnant or lactating females;
  2. Study participants with a history of neurological disease, such as epilepsy, intracranial hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, memory impairment, spinal cord compression, psychiatric disorders or any disease involving the central nervous system, or suspected central nervous system (CNS) metastasis;
  3. Presence of HIV, syphilis infection, active hepatitis B virus infection (HBV-DNA above detection limit or positive), or active hepatitis C virus infection (HCV-RNA positive);
  4. Current presence of any uncontrolled active infection, including but not limited to active tuberculosis study participants (as judged by the investigator);
  5. Known or suspected long-term active EBV infection, known history of HLH;
  6. The toxicities caused by previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE 5.0) ≤ Grade 1, except for alopecia and other tolerable events as judged by the investigator;
  7. Received autologous stem cell transplantation within 12 weeks before signing the informed consent form; Received allogeneic stem cell transplantation;
  8. Prior treatment targeting CD19 (unless the CD19 or CD20 target remains positive);
  9. Antineoplastic therapy, including but not limited to cytotoxic therapy, monoclonal antibodies or antibody conjugates, targeted therapy, radiotherapy, epigenetic therapy, or investigational drug therapy, or use of an invasive investigational medical device within 14 days or 5 half-lives (whichever is shorter) prior to cell infusion. Participants are eligible for the study regardless of the end date of radiotherapy if the radiation field covers ≤ 5% bone marrow reserve;
  10. Systemic corticosteroids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical corticosteroids;
  11. Vaccination with live attenuated vaccines, inactivated vaccines or RNA vaccines within 4 weeks prior to signing the informed consent form;
  12. Allergy or intolerance to CLD drugs, tocilizumab, or allergy to the components of CT1194D cell infusion preparation (dimethyl sulfoxide/DMSO); Or previous history of other severe allergies such as anaphylactic shock;
  13. Study participants with any of the following cardiac conditions:

  <!-- -->

  1. New York Heart Association (NYHA) Class III or IV heart failure;
  2. Myocardial infarction, coronary artery bypass grafting, or unstable angina 6 months prior to screening;
  3. History of clinically significant uncontrolled arrhythmia, such as ventricular arrhythmia;
  4. History of severe non-ischemic cardiomyopathy;
  5. Other cardiac disease that, in the opinion of the investigator, may jeopardize the health of the study participant due to participation in this clinical study; 14. Have other severe pulmonary disease that may endanger the life of the study participant as judged by the investigator; 15. Have a second primary malignancy requiring treatment or not in complete remission within the past 2 years, with the exception of successfully treated non-metastatic basal cell or squamous cell skin cancer, non-metastatic carcinoma in situ of the prostate, breast or cervical cancer, non-muscle invasive bladder cancer or thyroid cancer and other low-grade tumors; 16. Study participants with active autoimmune diseases, including but not limited to psoriasis, rheumatoid arthritis, inflammatory bowel disease and other diseases requiring long-term immunosuppressive therapy; 17. Major surgery within 2 weeks before signing the informed consent form, or planning to undergo major surgery during the study or within 4 weeks after the administration of study treatment (excluding cataract and other surgery under local anesthesia); 18. Inability or unwillingness of the participant to comply with the requirements of the study protocol as assessed by the investigator, or for other reasons unsuitable for participation in this clinical study.
* R/R B-ALL Inclusion Criteria：

  1. Pregnant or lactating females;
  2. Study participants with a history of neurological disorders, such as epilepsy, intracranial hemorrhage, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, memory impairment, spinal cord compression, psychiatric disorders or any disease involving the central nervous system, or active central nervous system (CNS) leukemia;
  3. Presence of HIV, syphilis infection, active hepatitis B virus infection (HBV-DNA above detection limit or positive), or active hepatitis C virus infection (HCV-RNA positive);
  4. Current presence of any uncontrolled active infection, including but not limited to active tuberculosis study participants (as judged by the investigator);
  5. Known or suspected long-term active EBV infection, known history of HLH;
  6. Presence of active systemic autoimmune disease;
  7. The toxicities caused by previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE V5.0) ≤ Grade 1, except for alopecia and other tolerable events as judged by the investigator;
  8. Study participants with solitary extramedullary lesions; Study participants with genetic syndromes associated with bone marrow failure states: such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome.
  9. Study participants who relapsed after treatment with drugs targeting CD19 and/or CD20 prior to screening and who are judged not to benefit by the investigator;
  10. Received autologous or allogeneic stem cell transplantation within 3 months before signing the informed consent form; Donor lymphocyte infusion (DLI) within 6 weeks;
  11. Active graft-versus-host disease (GVHD) of grade 2-4 within 4 weeks before signing the informed consent form;
  12. Antineoplastic therapy, including but not limited to cytotoxic therapy, monoclonal antibodies or antibody conjugates, targeted therapy, radiotherapy, epigenetic therapy, or investigational drug therapy, or use of an invasive investigational medical device within 14 days or 5 half-lives (whichever is shorter) prior to cell infusion. Participants are eligible for the study regardless of the end date of radiotherapy if the radiation field covers ≤ 5% bone marrow reserve;
  13. Systemic corticosteroids equivalent to > 15 mg/day prednisone within 3 days prior to cell infusion, except for topical corticosteroids;
  14. Vaccination with live attenuated vaccines, inactivated vaccines or RNA vaccines within 4 weeks prior to signing the informed consent form;
  15. Allergy or intolerance to CLD drugs, tocilizumab, or allergy to the components of CT1194D cell infusion preparation (dimethyl sulfoxide/DMSO); Or previous history of other severe allergies such as anaphylactic shock;
  16. Study participants with any of the following cardiac conditions:

  <!-- -->

  1. New York Heart Association (NYHA) Class III or IV heart failure;
  2. Myocardial infarction, coronary artery bypass grafting, or unstable angina 6 months prior to screening;
  3. History of clinically significant uncontrolled arrhythmia, such as ventricular arrhythmia;
  4. History of severe non-ischemic cardiomyopathy;
  5. Other cardiac disease that, in the opinion of the investigator, may jeopardize the health of the study participant due to participation in this clinical study; 17. Have other severe pulmonary disease that may endanger the life of the study participant as judged by the investigator; 18. Have a second primary malignancy requiring treatment or not in complete remission within the past 2 years, with the exception of successfully treated non-metastatic basal cell or squamous cell skin cancer, non-metastatic carcinoma in situ of the prostate, breast or cervical cancer, non-muscle invasive bladder cancer or thyroid cancer and other low-grade tumors; 19. Major surgery within 2 weeks before signing the informed consent form, or planning to undergo major surgery during the study or within 4 weeks after the administration of study treatment (excluding cataract and other surgery under local anesthesia); 20. After organ transplantation; 21. Inability or unwillingness of the participant to comply with the requirements of the study protocol as assessed by the investigator, or for other reasons unsuitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess the severity and incidence of DLTs, treatment-related adverse events (TRAE), and adverse events of special interest (AESI) after CT1194D infusion | 12 months after CT1194D infusion
MTD or dose range | Up to 28 days after CAR-T cells infusion
  To explore the maximum tolerated dose (MTD) or dose range of CT1194D

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Evaluate at 4, 8, 12 weeks and 6,9,12month after CAR-T infusion
Complete response rate (CRR) | 12 months after CT1194D infusion
Minimal Residual Disease Negative (MRD-) Proportion (R/R B-ALL) | 12 months after CT1194D infusion
Duration of response (DOR) | 12 months after CT1194D infusion
Time to response (TTR) | 12 months after CT1194D infusion
Time to complete response (TTCR) | 12 months after CT1194D infusion
Progression-free survival (PFS) | 12 months after CT1194D infusion
Overall Survival (OS) | 12 months after CT1194D infusion

CONTACTS AND LOCATIONS:
Locations (1):
- China Institute of Hematology and Blood Diseases Hospital, Tianjin, China